CLINICAL TRIAL: NCT07281495
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study With Open-Label Extension to Assess the Efficacy, Safety, and Pharmacokinetics of Subcutaneously Administered Taldefgrobep Alfa in Adults Living With Overweight and Obesity
Brief Title: Taldefgrobep Alfa in Adults With Overweight and Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV2000-202
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: myostatin; activin
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Taldefgrobep Alpha once weekly (Experimental)
  Interventions: Drug: Taldefgrobep Alfa
- Placebo once weekly (Placebo Comparator)
  Interventions: Drug: Placebo
- Taldefgrobep Alpha once every 4 weeks (Experimental)
  Interventions: Drug: Taldefgrobep Alfa
- Placebo once every 4 weeks (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Taldefgrobep Alfa — Subcutaneous injection administered once each week
  Other Names: BHV-2000
  Arms: Taldefgrobep Alpha once weekly
Drug: Placebo — Subcutaneous injection (matching placebo) administered once each week
  Arms: Placebo once weekly
Drug: Taldefgrobep Alfa — Subcutaneous injection administered once every 4 weeks
  Other Names: BHV-2000
  Arms: Taldefgrobep Alpha once every 4 weeks
Drug: Placebo — Subcutaneous injection (matching placebo) administered once every 4 weeks
  Arms: Placebo once every 4 weeks

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, multiple dose study to evaluate the efficacy, safety, and tolerability of taldefgrobep alfa in adults with overweight and obesity, with an open-label extension.

ELIGIBILITY:
Key Inclusion Criteria:

1. a. BMI > 30 kg/m2 and BMI < 42 kg/m2, OR b. BMI ≥ 27 kg/m2 and BMI <30 kg/m2 with at least one weight-related co-morbidity
2. History of at least one self-reported unsuccessful dietary effort to lose body weight.
3. Stable body weight and stable physical activity within 3 months prior to screening per participant self-report.
4. All participants must adhere to protocol contraception requirements

Key Exclusion Criteria:

1. History of diabetes, including individuals with a HbA1c of ≥ 6.5% at Screening
2. Non-ambulatory participants, defined as unable to take at least 10 steps independently.
3. Females currently pregnant or breastfeeding, or who intend to become pregnant or to breastfeed.
4. Participation in another investigational clinical trial while participating in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in total body weight from Baseline to Week 24 | Baseline to Week 24

SECONDARY OUTCOMES:
Percent change in total body fat mass from Baseline to Week 24 | Baseline to Week 24
Percent change in total body lean mass from Baseline to Week 24 | Baseline to Week 24
Number of participants with death, SAEs, AEs considered related to study drug, moderate and severe AEs, and Grade 3 to 4 laboratory abnormalities | Through week 24

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Site-001, Chula Vista, California
  - Site-014, Montclair, California
  - Site-011, Sacramento, California
  - Site-018, Tustin, California
  - Site-008, Palm Springs, Florida
  - Site-015, St. Petersburg, Florida
  - Site-007, Chicago, Illinois
  - Site-016, Indianapolis, Indiana
  - Site-010, Baton Rouge, Louisiana
  - Site-009, Metairie, Louisiana
  - Site-006, City of Saint Peters, Missouri
  - Site-003, Springfield, Missouri
  - Site-019, Monroe, North Carolina
  - Site-002, Fargo, North Dakota
  - Site-017, North Charleston, South Carolina
  - Site-005, Austin, Texas
  - Site-012, McKinney, Texas
  - Site-013, San Antonio, Texas
  - Site-004, Arlington, Virginia